CLINICAL TRIAL: NCT01095848
Title: A Phase I Study of Two Different Doses of the Subcutaneous Administration of an Immunotherapeutic Vaccine, DPX-0907 in Advanced Stage Patients With Ovarian, Breast or Prostate Cancer
Brief Title: A Phase I Safety Study of a Cancer Vaccine to Treat HLA-A2 Positive Advanced Stage Ovarian, Breast and Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunoVaccine Technologies, Inc. (IMV Inc.) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONC-DPX-0907-01
Record Dates: First submitted 2010-03-26; First posted 2010-03-30 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Ovarian Neoplasms; Breast Neoplasms; Prostatic Neoplasms
Keywords: vaccine; cancer; ovarian; breast; prostate; tumor; Immunotherapy
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.25ml dose DPX-0907 (Experimental): On each vaccination day the lyophilized antigen/adjuvant/liposome complex is re-suspended in the oil (Montanide 1SA51 VG) before injection. The vaccine is not an emulsion.
  Interventions: Biological: DPX-0907 consists of 7 tumor-specific HLA-A2-restricted peptides, a universal T Helper peptide, a polynucleotide adjuvant, a liposome and Montanide ISA51 VG
- 1ml dose DPX-0907 (Experimental): On each vaccination day the lyophilized antigen/adjuvant/liposome complex is re-suspended in the oil (Montanide 1SA51 VG) before injection. The vaccine is not an emulsion.
  Interventions: Biological: DPX-0907 consists of 7 tumor-specific HLA-A2-restricted peptides, a universal T Helper peptide, a polynucleotide adjuvant, a liposome and Montanide ISA51 VG

INTERVENTIONS:
Biological: DPX-0907 consists of 7 tumor-specific HLA-A2-restricted peptides, a universal T Helper peptide, a polynucleotide adjuvant, a liposome and Montanide ISA51 VG — Patients will receive three deep subcutaneous injections of the vaccine three weeks apart in the upper thigh region. Patients will be followed for up to 7 months.

SUMMARY:
To determine the safety and immunogenicity profile of two (2) different doses of the vaccine DPX-0907 to treat breast, ovarian and prostate cancer.

DETAILED DESCRIPTION:
Epithelial ovarian cancer has a high mortality rate even among those who obtain complete remission after surgery and chemotherapy. In prostate cancer, hormonal therapies including androgen ablation may control the disease for variable lengths of time but progression will invariably occur. There is also a high rate of relapse in breast cancer patients who have four or more positive axillary lymph nodes and in cases of resected metastatic disease. Immune therapies such as therapeutic vaccination may prolong remissions in these cancers.

Many different therapeutic vaccines have been evaluated in these diseases in phase 1, 2 and even phase 3 trials. Much has been learned about the principals of applying immune-based therapies and specifically the types of patients that may be most likely to mount an effective immune response. Cancer vaccines may have their greatest impact earlier in the disease course or in situations with minimal residual disease. Most recently an overall survival benefit was documented in prostate cancer patients with an immunotherapy based vaccine.

ImmunoVaccine Technologies Inc. (IVT) is developing a therapeutic vaccine against various solid cancers based on a patented vaccine delivery and enhancement platform. The antigens included in DPX-0907 were identified using an innovative antigen discovery platform to identify proprietary signature antigens actually presented on the surface of tumor cells and therefore capable of stimulating a cellular immune response in the patient. One or more of the peptide antigens are expected to be expressed in the types of tumors included in this trial. The peptide antigens proposed for DPX-0907 have been previously included in a phase I study in a different vaccine formulation at Duke University. No vaccine-induced autoimmune events were reported. These encouraging results suggest that the autoimmune potential of these cancer-specific peptide antigens is limited. IVT's DepoVax™ (DPX) lipid-based formulation was designed to enhance the speed, strength and duration of the cellular immune response. This formulation in combination with tumor targeting antigens has produced favorable safety and cellular immune responses in preclinical studies. These parameters will be studied in this phase I trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage III or IV ovarian cancer who have completed a course of platinin-based cytotoxic therapy after debulking surgery with evidence of a complete or partial response by radiological imaging. Patients with metastatic ovarian cancer who have stable disease for greater than 3 months after completion of first-line therapy.
* Patients with stage IV breast cancer who have received at least 1 course of hormonal or cytotoxic therapy for metastatic cancer. Patients must be off cytotoxic therapy with stable disease or better for 3 months or greater duration. Patients may have stable disease and still be on hormonal therapy.
* Patients with prostate cancer who have failed at least 1 course of an accepted hormonal therapy. Specifically prostate cancer patients must have castrate testosterone levels (< 50 ng/dl) and 2 PSA values higher than the previously documented baseline at least 3 weeks apart or evidence of increases in measurable disease. These patients may have received previous courses of cytotoxic chemotherapy although chemotherapy naïve patients who are deemed not good candidates or who have refused cytotoxic therapy will be eligible. These patients may remain on anti-androgen therapy during the trial. Patients with evidence of progressive bone or other metastases are acceptable.
* At least 8 weeks since previous courses of an investigational biologic therapy (i.e. cancer vaccine) including active or passive immunotherapy.
* At least 30 days since localized surgery or radiotherapy.
* At least 30 days since initiation of a biphosphonate treatment.
* HLA A2 haplotype.

Exclusion Criteria:

* History of autoimmune disease, such as inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis. Patients with a remote history (greater than five years) of thyroiditis are not excluded.
* Presence of an acute infection requiring antibiotics within 4 weeks of study entry or a chronic infection such as: urinary tract infection, HIV, or antigen positive viral hepatitis.
* Previously resected brain metastases unless a CT or MRI scan of the brain shows no metastasis within 1 month of receiving DPX-0907.
* Concurrent (within the last 5 years) second malignancy other than non-melanoma skin cancer, cervical carcinoma in situ, or controlled bladder cancer.
* Acute or chronic skin disorders that will interfere with subcutaneous injection of the vaccine or subsequent assessment of potential skin reactions.
* Serious intercurrent chronic or acute illness, such as cardiac disease (NYHA class III or IV) or hepatic disease.
* Steroid therapy or other immunosuppressives, such as azathioprine or cyclosporin A, unless steroids are discontinued 6 weeks prior to study.
* Allergies to any component of the vaccine.
* Inability to gain venous access.
* Previous splenectomy.
* Previous lymphadenectomy in both inguinal regions.
* Pregnant or nursing mothers.
* Medical or psychological impediment or active drug or alcohol use that might preclude protocol compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-03; Primary Completion 2011-04 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To determine the safety profile of two different doses of subcutaneously administered DPX-0907. Safety assessments will be based on reported adverse events and the results of vital sign measurements, physical examinations, and clinical laboratory tests. | On each vaccination day, 30 days after last vaccination and every month during the 6 month follow-up period

SECONDARY OUTCOMES:
To determine the levels of CMI (cell mediated immunity) to the 7 cancer epitopes induced by vaccination with DPX-0907 | On each vaccination day, 30 days after last vaccination
To establish a recommended dose based on safety and immune response for phase 2 studies. | On each vaccination day, 30 days after last vaccination and every month during the 6 month follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morse, MD, Study Chair — Duke University
Locations (5):
- United States (5):
  - Rush University Medical Center, Chicago, Illinois
  - Roswell Park Cancer Institute, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Mary Crowley Cancer Research Center, Dallas, Texas

REFERENCES:
- [Result] Berinstein NL, Karkada M, Morse MA, Nemunaitis JJ, Chatta G, Kaufman H, Odunsi K, Nigam R, Sammatur L, MacDonald LD, Weir GM, Stanford MM, Mansour M. First-in-man application of a novel therapeutic cancer vaccine formulation with the capacity to induce multi-functional T cell responses in ovarian, breast and prostate cancer patients. J Transl Med. 2012 Aug 3;10:156. doi: 10.1186/1479-5876-10-156. PMID 22862954